CLINICAL TRIAL: NCT05041335
Title: Wet Heparinized Suction: A Novel Technique to Enhance Tissue Acquisition for Endoscopic Ultrasound Guided Fine Needle Biopsy (EUS-FNB) of Solid Abdominal Masses: A Randomized Prospective Trial
Brief Title: Wet Heparinized Suction for Abdominal Cancer
Acronym: EUS Heparin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MCC-21926
Record Dates: First submitted 2021-02-15; First posted 2021-09-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cancer of Pancreas; Cancer of Stomach; Cancer of Esophagus; Cancer of Liver; Cancer
Keywords: cancer; esophagus; stomach; gastric; pancreas; biliary; bile; bile duct; liver; hepatic
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The control group will have 21 patients and the group receiving heparin will have 21 patients; the randomization is 1:1:1:1; heparin and microsieve, heparin and no microsieve, no heparin and microsieve and no heparin and no microsieve. Forty two subjects will be enrolled at UH for a total of 42 subjects.
Who Masked: Participant, Care Provider, Investigator
Masking Description: These needle preparations will be wrapped in non-transparent 2-inch tape to hide the appearance of the injectate agent. The needle is prepared by removing the stylet and flushing with the selected substance. The PI/Co-I will then flush the needle with the selected substance until drops of the liquid are seen exiting the needle tip. Those randomized to have the needle flushed with heparin will be termed "dry heparin" and will be flushed with 500 U heparin USP per 10 mL. Those who randomize not to receive heparin, the needle will be flushed with saline. The device shall then be placed into the linear echoendoscope and the FNB will be performed. The PI is blinded to heparin vs. no heparin only. Randomization to the microsieve vs. not is apparent to the PI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Heparin and microsieve (Experimental): The needle will be prepped with 500 U heparin USP per 10 mL to coat the inside of the needle. The provider will expel the tissue onto the microsieve
  Interventions: Other: wet heparinzed suction; Other: Microsieve
- Heparin and no microsieve (Experimental): The needle will be prepped with 500 U heparin USP per 10 mL to coat the inside of the needle. The provider will expel the tissue into formalin
  Interventions: Other: wet heparinzed suction; Other: No microsieve
- No heparin and microsieve (Experimental): The needle not be prepped. The provider will expel the tissue onto the microsieve
  Interventions: Other: Microsieve; Other: No heparin flush
- No heparina nd no microsieve (Active Comparator): The needle not be prepped. The provider will expel the tissue into formalin
  Interventions: Other: No heparin flush; Other: No microsieve

INTERVENTIONS:
Other: wet heparinzed suction — Needle flushed with 5000 Units in 10mL of heparin
  Arms: Heparin and microsieve; Heparin and no microsieve
Other: Microsieve — A microsieve used for tissue preparation
  Arms: Heparin and microsieve; No heparin and microsieve
Other: No heparin flush — The needle not prepped
  Arms: No heparin and microsieve; No heparina nd no microsieve
Other: No microsieve — The tissue is placed into formalin
  Arms: Heparin and no microsieve; No heparina nd no microsieve

SUMMARY:
The purpose of this research is to compare the amount and quality of tissue obtained by EUS-FNB when the device is flushed with an anticoagulant or "blood thinner" vs. saline a salt water solution as well as the use of a microsieve in order for the doctor to look at the tissue to check the acceptability of the specimens before sending for analysis.

You will be randomly assigned (like a flip of a coin) to have either the blood thinner or the salt water solution placed within the needle being used to sample your abdominal tumor and to have either a sieve used or not.

You will be one of 42 participants enrolled in this data collection study which includes 1 sites in the United States.

DETAILED DESCRIPTION:
Since its inception in the early 1990's, endoscopic ultrasound with fine needle aspiration (EUS-FNA) has developed into an important method for obtaining diagnostically accuracy for gastrointestinal, and extra-luminal pathology [1,2]. Present society guidelines by both the European Society of Gastrointestinal Endoscopy (ESGE) and American Society of Gastrointestinal Endoscopy (ASGE) have estimated an overall 60-90% diagnostic accuracy of EUS-FNA [2,3]. However, this accuracy is dependent upon determination of adequacy by expert gastrointestinal pathologists, which may not be available at all centers [4-6].

New developments in needle technology has led to development of "core needles", which can allow for acquisition of a tissue specimen with intact tissue architecture and therefore more ability for immunohistochemical staining (IHC). When evaluating pancreatic lesions, FNB needles have demonstrated 81-100% technical success and up to 94.7% diagnostic accuracy [18-21]. Overall, EUS-FNB appears to be a promising addition to EUS guided tissue acquisition, which has the potential of leading to improved diagnostic accuracy.

As an additional means for optimizing EUS-FNB, heparin has been described and studied in the past. The study investigators have been using heparin to prime the wet suction needle to prevent formation of clot in the needle which produces "blood noodles" in the specimen that can interfere with tissue processing and interpretation. There are previous data demonstrating that heparin priming of the needle may also increase yield [22]. The study investigators have demonstrated that use of a heparin primed needle does not interfere with cytology, histology or immunohistochemical analysis, and may ease stylet handling [23]. Also, the study investigators have directly validated the use of heparin for EUS-guided liver biopsies (EUS-LB) demonstrating improvement in the size and number of histologic fragments obtained from EUS-guided biopsy [24-25]. Given this information, heparin flush is actively used and readily available, in EUS-guided biopsies here at UH.

Rapid onsite cytological evaluation (ROSE) has been used to make an immediate assessment of tissue adequacy during the EUS-FNA procedure, as well as to deliver a rapid pathological diagnosis during the EUS session. ROSE has been shown to increase the yield while having the potential of decreasing the number of needle passes required. However, ROSE is not available at many EUS centers. It would be advantageous to predict adequacy of a needle biopsy specimen without having to rely on ROSE.

In standard EUS-FNA practice, part of the biopsy specimens is used to prepare a smear that can be examined microscopically. The remainder of the specimen processed by the laboratory for "cell block" analysis. Microscopic examination of the smears and the cell-block are done by the pathologist to arrive at a final diagnosis.

The study investigators have developed a new technique of specimen enrichment using a "microsieve device". In this technique, a small microsieve collects the larger tissue fragments, while single cells and small cell clusters wash through the microsieve. Visible tissue fragments or cores likely represent a macroscopic representation of adequacy of tissue, and could theoretically supplant ROSE in providing an on-site determination of adequacy.

In the course of this study, the study investigators will collect the larger fragments as well as the wash-through and examine each separately.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year
* Non-pregnant Patients
* Patients with the presence of a solid abdominal mass as seen on diagnostic imaging [ie. ultrasound (US), computer tomography (CT) or magnetic resonance imaging (MRI)] scheduled to undergo EUS examination OR Patients who underwent a prior EUS-FNA/FNB for solid pancreatic mass and did not receive a conclusive diagnosis
* Patients with platelet count > 50,000
* Patients with International Normalized Ratio (INR) < 1.5

Exclusion Criteria:

* Age < 18 years
* Pregnant Patients
* Patients who cannot consent for themselves
* Patients with anticoagulants or anti-platelet agents (excluding aspirin) within the last 7-10 days
* Patients with cystic abdominal masses
* Patients with a platelet count < 50,000
* Patients with an INR > 1.5
* Patients with a heparin or porcine allergy
* Patients with prior heparin induced thrombocytopenia (HIT)
* Patient's with religious aversion to porcine-containing products

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-01-12 (Estimated)

PRIMARY OUTCOMES:
Aggregate specimen length (ASL) | immediately after the intervention/procedure/surgery
  sum length of all pieces of tissue obtained from EUS-FNB

SECONDARY OUTCOMES:
Length of the longest piece (LLP) | immediately after the intervention/procedure/surgery
  total length of the longest tissue piece
Mean number of small pieces | immediately after the intervention/procedure/surgery
  defined by pieces measuring <4 mm in length
Mean number of medium pieces | immediately after the intervention/procedure/surgery
  defined by pieces measuring 5-8 mm in length
Means number of long pieces | immediately after the intervention/procedure/surgery
  defined by pieces measuring >9 mm in length
Histology adequacy score | immediately after the intervention/procedure/surgery
  Histology adequacy score, defined as 1, a pathologist can make a clinical diagnosis using the tissue obtained or 0 a pathologist cannot make a clinical diagnosis using the tissue obtained
Presence of a visible core specimen | immediately after the intervention/procedure/surgery
  defined as 1, visible tissue seen by the endoscopist at the time of tissue preparation or 0 no visible tissue seen by the endoscopist at the time of tissue preparation
Presence of visible clots in specimen | immediately after the intervention/procedure/surgery
  defined as 1, visible clots seen by the endoscopist at the time of tissue preparation or 0 visible clots seen by the endoscopist at the time of tissue preparation
Mean blood clot score during histology | immediately after the intervention/procedure/surgery
  Defined as (0: Nearly absent of red blood cells (RBC), 1+: Monolayer of RBC, no cluster formation, 2+: Aggregates of RBC present, < x40 high power field, 3+: Aggregates of RBC present, > x40 high power field).
Adequacy of diagnosis | immediately after the intervention/procedure/surgery
  based upon fluid washed out from the microsieve tissue sample defined by Smears with relatively abundant and well-visualized lesional material.

CONTACTS AND LOCATIONS:
Overall Officials: Shaffer Mok, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vilmann P, Jacobsen GK, Henriksen FW, Hancke S. Endoscopic ultrasonography with guided fine needle aspiration biopsy in pancreatic disease. Gastrointest Endosc. 1992 Mar-Apr;38(2):172-3. doi: 10.1016/s0016-5107(92)70385-x. No abstract available. PMID 1568614
- [Background] Dumonceau JM, Deprez PH, Jenssen C, Iglesias-Garcia J, Larghi A, Vanbiervliet G, Aithal GP, Arcidiacono PG, Bastos P, Carrara S, Czako L, Fernandez-Esparrach G, Fockens P, Gines A, Havre RF, Hassan C, Vilmann P, van Hooft JE, Polkowski M. Indications, results, and clinical impact of endoscopic ultrasound (EUS)-guided sampling in gastroenterology: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline - Updated January 2017. Endoscopy. 2017 Jul;49(7):695-714. doi: 10.1055/s-0043-109021. Epub 2017 May 16. PMID 28511234
- [Background] Hebert-Magee S, Bae S, Varadarajulu S, Ramesh J, Frost AR, Eloubeidi MA, Eltoum IA. The presence of a cytopathologist increases the diagnostic accuracy of endoscopic ultrasound-guided fine needle aspiration cytology for pancreatic adenocarcinoma: a meta-analysis. Cytopathology. 2013 Jun;24(3):159-71. doi: 10.1111/cyt.12071. PMID 23711182
- [Background] Iglesias-Garcia J, Dominguez-Munoz JE, Abdulkader I, Larino-Noia J, Eugenyeva E, Lozano-Leon A, Forteza-Vila J. Influence of on-site cytopathology evaluation on the diagnostic accuracy of endoscopic ultrasound-guided fine needle aspiration (EUS-FNA) of solid pancreatic masses. Am J Gastroenterol. 2011 Sep;106(9):1705-10. doi: 10.1038/ajg.2011.119. Epub 2011 Apr 12. PMID 21483464
- [Background] Eloubeidi MA, Tamhane A, Jhala N, Chhieng D, Jhala D, Crowe DR, Eltoum IA. Agreement between rapid onsite and final cytologic interpretations of EUS-guided FNA specimens: implications for the endosonographer and patient management. Am J Gastroenterol. 2006 Dec;101(12):2841-7. doi: 10.1111/j.1572-0241.2006.00852.x. Epub 2006 Oct 6. PMID 17026562
- [Background] Jhala NC, Jhala DN, Chhieng DC, Eloubeidi MA, Eltoum IA. Endoscopic ultrasound-guided fine-needle aspiration. A cytopathologist's perspective. Am J Clin Pathol. 2003 Sep;120(3):351-67. doi: 10.1309/MFRF-J0XY-JLN8-NVDP. PMID 14502798
- [Background] Itoi T, Itokawa F, Sofuni A, Nakamura K, Tsuchida A, Yamao K, Kawai T, Moriyasu F. Puncture of solid pancreatic tumors guided by endoscopic ultrasonography: a pilot study series comparing Trucut and 19-gauge and 22-gauge aspiration needles. Endoscopy. 2005 Apr;37(4):362-6. doi: 10.1055/s-2004-826156. PMID 15824948
- [Background] Larghi A, Capurso G, Carnuccio A, Ricci R, Alfieri S, Galasso D, Lugli F, Bianchi A, Panzuto F, De Marinis L, Falconi M, Delle Fave G, Doglietto GB, Costamagna G, Rindi G. Ki-67 grading of nonfunctioning pancreatic neuroendocrine tumors on histologic samples obtained by EUS-guided fine-needle tissue acquisition: a prospective study. Gastrointest Endosc. 2012 Sep;76(3):570-7. doi: 10.1016/j.gie.2012.04.477. PMID 22898415
- [Background] Iwashita T, Yasuda I, Doi S, Ando N, Nakashima M, Adachi S, Hirose Y, Mukai T, Iwata K, Tomita E, Itoi T, Moriwaki H. Use of samples from endoscopic ultrasound-guided 19-gauge fine-needle aspiration in diagnosis of autoimmune pancreatitis. Clin Gastroenterol Hepatol. 2012 Mar;10(3):316-22. doi: 10.1016/j.cgh.2011.09.032. Epub 2011 Oct 20. PMID 22019795
- [Background] Diehl DL, Mok SRS, Khara HS, Johal AS, Kirchner HL, Lin F. Heparin priming of EUS-FNA needles does not adversely affect tissue cytology or immunohistochemical staining. Endosc Int Open. 2018 Mar;6(3):E356-E362. doi: 10.1055/s-0043-121880. Epub 2018 Mar 7. PMID 29527558
- [Background] Kasugai H, Yamamoto R, Tatsuta M, Okano Y, Okuda S, Kishigami Y, Kitamura T, Wada A, Tamura H. Value of heparinized fine-needle aspiration biopsy in liver malignancy. AJR Am J Roentgenol. 1985 Feb;144(2):243-4. doi: 10.2214/ajr.144.2.243. PMID 2981458
- [Background] Mok SRS, Diehl DL, Johal AS, Khara HS, Confer BD, Mudireddy PR, Kirchner HL, Chen ZE. A prospective pilot comparison of wet and dry heparinized suction for EUS-guided liver biopsy (with videos). Gastrointest Endosc. 2018 Dec;88(6):919-925. doi: 10.1016/j.gie.2018.07.036. Epub 2018 Aug 16. PMID 30120956
- [Background] Attam R, Arain MA, Bloechl SJ, Trikudanathan G, Munigala S, Bakman Y, Singh M, Wallace T, Henderson JB, Catalano MF, Guda NM. "Wet suction technique (WEST)": a novel way to enhance the quality of EUS-FNA aspirate. Results of a prospective, single-blind, randomized, controlled trial using a 22-gauge needle for EUS-FNA of solid lesions. Gastrointest Endosc. 2015;81(6):1401-7. doi: 10.1016/j.gie.2014.11.023. Epub 2015 Feb 27. PMID 25733127
- [Background] Schulman AR, Thompson CC, Odze R, Chan WW, Ryou M. Optimizing EUS-guided liver biopsy sampling: comprehensive assessment of needle types and tissue acquisition techniques. Gastrointest Endosc. 2017 Feb;85(2):419-426. doi: 10.1016/j.gie.2016.07.065. Epub 2016 Aug 13. PMID 27530070
- [Background] Thomas T, Kaye PV, Ragunath K, Aithal G. Efficacy, safety, and predictive factors for a positive yield of EUS-guided Trucut biopsy: a large tertiary referral center experience. Am J Gastroenterol. 2009 Mar;104(3):584-91. doi: 10.1038/ajg.2008.97. Epub 2009 Feb 10. PMID 19262518
- [Background] Wahnschaffe U, Ullrich R, Mayerle J, Lerch MM, Zeitz M, Faiss S. EUS-guided Trucut needle biopsies as first-line diagnostic method for patients with intestinal or extraintestinal mass lesions. Surg Endosc. 2009 Oct;23(10):2351-5. doi: 10.1007/s00464-009-0345-2. Epub 2009 Mar 5. PMID 19263153
- [Background] Sey MS, Al-Haddad M, Imperiale TF, McGreevy K, Lin J, DeWitt JM. EUS-guided liver biopsy for parenchymal disease: a comparison of diagnostic yield between two core biopsy needles. Gastrointest Endosc. 2016 Feb;83(2):347-52. doi: 10.1016/j.gie.2015.08.012. Epub 2015 Aug 13. PMID 26278654
- [Background] Gleeson FC, Clayton AC, Zhang L, Clain JE, Gores GJ, Rajan E, Smyrk TC, Topazian MD, Wang KK, Wiersema MJ, Levy MJ. Adequacy of endoscopic ultrasound core needle biopsy specimen of nonmalignant hepatic parenchymal disease. Clin Gastroenterol Hepatol. 2008 Dec;6(12):1437-40. doi: 10.1016/j.cgh.2008.07.015. Epub 2008 Jul 26. PMID 19081532
- [Background] Nieto J, Khaleel H, Challita Y, Jimenez M, Baron TH, Walters L, Hathaway K, Patel K, Lankarani A, Herman M, Holloman D, Saab S. EUS-guided fine-needle core liver biopsy sampling using a novel 19-gauge needle with modified 1-pass, 1 actuation wet suction technique. Gastrointest Endosc. 2018 Feb;87(2):469-475. doi: 10.1016/j.gie.2017.05.013. Epub 2017 May 24. PMID 28551024
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Burlingame OO, Kesse KO, Silverman SG, Cibas ES. On-site adequacy evaluations performed by cytotechnologists: correlation with final interpretations of 5241 image-guided fine-needle aspiration biopsies. Cancer Cytopathol. 2012 Jun 25;120(3):177-84. doi: 10.1002/cncy.20184. Epub 2011 Aug 31. PMID 21882357
- [Background] Mok SRS, Diehl DL, Johal AS, Khara HS, Confer BD, Mudireddy PR, Kovach AH, Diehl MM, Kirchner HL, Chen ZE. Endoscopic ultrasound-guided biopsy in chronic liver disease: a randomized comparison of 19-G FNA and 22-G FNB needles. Endosc Int Open. 2019 Jan;7(1):E62-E71. doi: 10.1055/a-0655-7462. Epub 2019 Jan 4. PMID 30648141
- [Background] Mok SRS, Diehl DL. The Role of EUS in Liver Biopsy. Curr Gastroenterol Rep. 2019 Jan 31;21(2):6. doi: 10.1007/s11894-019-0675-8. PMID 30706151